CLINICAL TRIAL: NCT05260723
Title: RISE - A Pilot Study to Reduce Sitting Time Among Breast Cancer Survivors
Brief Title: RISE - Reduce Sitting Time Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheri Hartman, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PILOT 171548
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Sedentary Behavior; Sedentary Time; Breast Cancer
Keywords: Physical Function; Cognitive Function; Quality of Life
MeSH Terms: conditions — Sedentary Behavior; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sit Less (Experimental): The primary goal of the Sit Less arm is to reduce the total amount of time spent sitting each day and break up prolonged bouts of sitting.
  Interventions: Behavioral: Behavioral: Sit Less

INTERVENTIONS:
Behavioral: Behavioral: Sit Less — The Sit Less arm uses habit formation, social cognitive theory, and motivational interviewing techniques to support behavior change and includes: 1) 7 health coaching sessions to set personalized goals and review progress; 2) wearing an activPAL (thigh worn accelerometer that measures sitting time); 3) intervention tools to support behavior change (e.g., standing desk, wrist worn monitor).

SUMMARY:
This 3-month study will test whether a program to reduce sitting time, for breast cancer survivors experiencing some physical limitations, can improve their physical function and other important aspects of quality of life.

DETAILED DESCRIPTION:
Many cancer survivors experience long-term physical problems following their cancer treatments and can often seem much older than same age peers who were never treated for cancer. This is known as accelerated aging. One way to improve accelerated aging is to increase moderate to vigorous intensity exercise; however, for many cancer survivors, especially those with physical limitations, increasing exercise levels is not possible. Another potential way to improve accelerated aging may be to decrease the amount of time spent sitting. Long periods of sitting are related to many physical and health problems. Cancer survivors spend more than 9 hours a day sitting and often increase the amount they sit after their cancer treatments. This study could help identify realistic intervention targets for many cancer survivors and be used to guide recommendations for improving physical function and quality of life after cancer.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivors (stages I-IV) at least 1 year post active treatment (e.g., chemotherapy, radiotherapy)
* Breast cancer was treated with chemotherapy, radiation, immunotherapy, and/or endocrine therapy
* self-report difficulties with physical function
* self-report low levels of moderate to vigorous physical activity
* self-report high levels of sitting time

Exclusion Criteria:

* medical condition that interferes with ability to safely stand or stay balanced
* other cancer diagnoses that occurred after their breast cancer diagnosis
* Stage IV breast cancer with brain metastases or less than 12 months life-expectancy
* unable to commit to a 3-month study

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-05-07 (Actual)

PRIMARY OUTCOMES:
Retention rate of enrolled participants | 3 months
  Percent of participants returning for the 3 month measures

SECONDARY OUTCOMES:
4 meter walk test | 3 months
  Measure of physical functioning
30-second Sit-to-Stand Test | 3 months
  Measure of physical functioning
Timed Up and Go (TUG) | 3 months
  Measure of physical functioning
Patient Reported Measurement Information System - Physical Function | 3 months
  Measure of Self-Report Physical Function, standardized T-score, higher scores indicated better functioning

CONTACTS AND LOCATIONS:
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States